CLINICAL TRIAL: NCT05665140
Title: Phase II Trial for Newly Diagnosed Low-risk Multiple Myeloma Patients Comparing 6 Cycles of Isatuximab With Lenalidomide/Bortezomib/Dexamethasone (I-VRD) Compared to 3 Cycles of I-VRD Followed by One Cycle of High-dose Therapy and Both Arms Followed by Maintenance Therapy With I-R.
Brief Title: Expression-linked and R-ISS-adapted Stratification for First Line Therapy in Multiple Myeloma Patients
Acronym: ELIAS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hopsital Schleswig Holstein Campus Lübeck (Other)
Responsible Party: Principal Investigator, Cyrus Khandanpour, Associate Professor and Deputy Director of Department of Haematology and Oncoloy, University Hopsital Schleswig Holstein Campus Lübeck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UZL22_01; 2022-500453-16-00 (Other: EU-CT-Number (CTIS))
Record Dates: First submitted 2022-11-28; First posted 2022-12-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Newly Diagnosed Multiple Myeloma
MeSH Terms: interventions — isatuximab; Lenalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Control) (Active Comparator): Three cycles of induction (isatuximab, bortezomib, lenalidomide, dexamethasone, I-VRD), followed by standard of care therapy (e.g. stem cell mobilization, and apheresis with a subsequent high-dose melphalan and autologous stem cell transfusion).
  Both groups will receive subsequently an isatuximab- and lenalidomide-based maintenance therapy.
  Interventions: Drug: Isatuximab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone; Other: autologous stem cell transplant
- Arm B (Experimental) (Experimental): Three cycles of induction (I-VRD), stem cell mobilization, and apheresis followed by three cycles of consolidation (I-VRD).
  Both groups will receive subsequently an isatuximab- and lenalidomide-based maintenance therapy.
  Interventions: Drug: Isatuximab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Isatuximab — i.v. Induction Phase (Arm A and B): Induction Cycle 1 10 mg/kg D 1, 8, 15, 22, 29. Induction Cycle 2-3 10 mg/kg D 1, 15, 29 Consolidation Phase (Arm B): Consolidation Cycle 1-3 10 mg/kg D 1, 15, 29 Maintenance Phase (Arm A and B): Maintenance Cycle 1 and subsequent cycles 10 mg/kg D 1, 15, 29
  Other Names: Sarclisa®
Drug: Lenalidomide — hard capsule for oral use. Induction Phase (Arm A and B): Induction Cycle 1-3 25 mg D1-14, 20-35. Consolidation Phase (Arm B): Consolidation Cycle 1-3 25 mg D1-14, 20-35. Maintenance Phase (Arm A and B): Maintenance Cycle 1-2 10 mg D1-28. Maintenance Cycle 3 and subsequent cycles 15 mg D1-28 if tolerable
  Other Names: Lenalidomid®
Drug: Bortezomib — s.c. injection. Induction Phase (Arm A and B): Induction Cycle 1-3 1,3 mg/m² D1, 4, 8, 11, 22, 25, 29, 32. Consolidation Phase (Arm B): Consolidation Cycle 1-3 1,3 mg/m² D1, 4, 8, 11, 22, 25, 29, 32
  Other Names: Velcade®
Drug: Dexamethasone — orally and i.v. Induction Phase (Arm A and B): Induction Cycle 1 20 mg p.o. D 1-2, 4-5, 8-9, 11-12, 15; 22-23, 25-26, 29-30, 32-33; 20 mg i.v. D1, 8, 15, 22 and 29. Induction Cycles 2 and 3 20 mg p.o. D 1-2, 4-5, 8-9, 11-12, 15; 22-23, 25-26, 29-30, 32-33; 20 mg i.v. D1, 15 and 29. Consolidation Phase (Arm B): Consolidation Cycle 1-3 20 mg p.o. on D 1-2, 4-5, 8-9, 11-12, 15; 22-23, 25-26, 29-30, 32-33; 20 mg i.v. on D1, 15 and 29
Other: autologous stem cell transplant — autologous stem cell transplant
  Arms: Arm A (Control)

SUMMARY:
Multiple myeloma (MM) is a malignant disease of the BM characterized by clonal expansion of plasma cells. Current guidelines recommend that newly diagnosed transplant-eligible patients with multiple myeloma (NDMMTE) shall undergo several cycles of induction, followed by one or two cycles high-dose melphalan followed by autologous stem cell transfusion (ASCT). Currently, induction therapy schemes usually consist of an immunomodulator (thalidomide or lenalidomide), a transmembrane glycoprotein CD38 targeting antibody, a proteasome inhibitor, and dexamethasone. The induction therapy is then followed by stem cell mobilization and subsequently one or two cycles of high-dose melphalan-chemotherapy based on the initial cytogenetic findings of the malignant plasma cells and the initial stage of the disease. Essentially, all NDMMTE patients undergo at least one cycle of high-dose chemotherapy, which is associated with high morbidity including acute toxicities like cytopenia, infection, and long-term effects such as myelodysplastic disease (MDS) and secondary malignancies and rarely death.

Based on preliminary data and published reports, exposure to high-doses of the genotoxic agent melphalan might render the residual malignant myeloma cells into more aggressive clones, accelerating relapse by potentially altering stroma. Finally, exposure to melphalan is well known to increase the possibility of secondary malignant disease development. In MM patients, high-dose melphalan therapy improves OS and PFS if patients from all risk groups are taken in consideration. Yet, it remains to be answered, whether also low risk patients have an additional benefit from high-dose melphalan therapy or whether for these patients, a less toxic regime would be similarly sufficient with regard to PFS and OS. The challenging question will be whether the effect of melphalan on initial disease control might be outpaced by the negative effects as described above. Hence, the sponsor will explore whether treatment with high-dose melphalan might represent an overtreatment for certain subpopulation myeloma patients. These patients might be adequately treated without need of high-dose melphalan as part of the first line treatment. The sponsor, therefore, proposes to use a personalized approach to evaluate whether patients with a low-risk profile and with a gene expression profile indicating a standard risk of relapse might be sufficiently treated with an intensified induction course without subsequent upfront high-dose melphalan chemotherapy.

DETAILED DESCRIPTION:
Multiple myeloma is a malignant disease of the BM characterized by clonal expansion of plasma cells. Current guidelines recommend that newly diagnosed transplant-eligible patients with multiple myeloma (NDMMTE) shall undergo several cycles of induction, followed by one or two cycles high-dose melphalan followed by autologous stem cell transfusion (ASCT). With the introduction of new drugs, the prognosis of multiple myeloma patients has considerably improved over time. Currently, induction therapy schemes usually consist of an immunomodulator (thalidomide or lenalidomide), a CD38 targeting antibody, a proteasome inhibitor, and dexamethasone. The induction therapy is then followed by stem cell mobilization and subsequently one or two cycles of high-dose melphalan-chemotherapy based on the initial cytogenetic findings of the malignant plasma cells and the initial stage of the disease. Current guidelines recommend two cycles of high-dose melphalan therapy followed by autologous stem cell transplantation in case of the following initial findings: presence of cytogenetic: (4;14), (14;16), (14;20) translocations or deletion 17p (del 17p), determined by fluorescence in situ hybridization (FISH). In addition, initial stage of R-ISS stage III leads also to the recommendation of two rounds of high-dose melphalan. Furthermore, if the patient does not achieve partial response as described by International Myeloma Working Group (IMWG) recommendations after the first cycles of high-dose melphalan, a second cycle of high-dose melphalan therapy should be administered. Later, patients treated outside clinical trials receive either 2-3 cycles of consolidation therapy and finally take lenalidomide (usually 10 or 15 mg on a daily basis) or proceed directly to a lenalidomide based maintenance therapy till progression or intolerable toxicity. Essentially, all NDMMTE patients undergo at least one cycle of high-dose chemotherapy, which is associated with high morbidity including acute toxicities like cytopenia, infection, and long-term effects such as myelodysplastic disease (MDS) and secondary malignancies and rarely death.

Based on preliminary data and published reports, exposure to high-doses of the genotoxic agent melphalan might render the residual malignant myeloma cells into more aggressive clones, accelerating relapse by potentially altering stroma. Finally, exposure to melphalan is well known to increase the possibility of secondary malignant disease development. In MM patients, high-dose melphalan therapy improves OS and PFS if patients from all risk groups are taken in consideration. Yet, it remains to be answered, whether also low risk patients have an additional benefit from high-dose melphalan therapy or whether for these patients, a less toxic regime would be similarly sufficient with regard to PFS and OS. The challenging question will be whether the effect of melphalan on initial disease control might be outpaced by the negative effects as described above. Hence, the sponsor will explore whether treatment with high-dose melphalan might represent an overtreatment for certain subpopulation myeloma patients. These patients might be adequately treated without need of high-dose melphalan as part of the first line treatment. We, therefore, propose to use a personalized approach to evaluate whether patients with a low-risk profile (R-ISS stage I, characterized by low tumor burden and absence of adverse cytogenetic findings or elevated LDH) and with a gene expression profile indicating a standard risk of relapse (please see below) might be sufficiently treated with an intensified induction course without subsequent upfront high-dose melphalan chemotherapy.

Personalized therapy can be achieved by considering gene expression analysis of the malignant BM cells together with the diagnostic work-up. We have a standardized CE-certified gene expression array, the MMprofilerTM, allowing accurate prediction of high-risk disease based on the SKY92 risk signature, calculating a risk score based on the expression of 92 genes from the malignant plasma cells. Its prognostic superiority has been analyzed in multiple retrospective analyses, totaling over 3,000 MM patients. This enables us to better define the aggressiveness of the disease and NDMMTE patient's 'individual' risk for disease progression within this research initiative and to define appropriate clinical strategies.

As an ultimate goal of this study, the sponsor aims to combine the outcome of gene expression array with the revised international staging system (R-ISS) to achieve a more personalized treatment. For patients with R-ISS stage I and the absence of high-risk disease as determined by the SKY92 signature (GEP-SR), the sponsor proposes a therapeutic approach without a requirement for high-dose chemotherapy as part of first-line therapy. This study would provide personalized treatment for myeloma patients, which could dramatically reduce toxicity, cost of therapy and lower the probability to develop a malignant clone (by about 25%) in all NDMMTE, and simultaneously improving the outcome of overall survival (OS) and progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed, untreated, symptomatic, documented myeloma (according to the revised Hypercalcaemia, renal dysfunction, anaemia and bone lesions (CRAB) criteria 2014, see Appendix 1) with clonal bone marrow (BM) plasma cells ≥10% or biopsy-proven osseous or extramedullary plasmacytoma and any one or more of the following myeloma defining events: I. Hypercalcemia: serum calcium >0,25 mmol/L (>1 mg/dl) higher than the upper limit of normal or >2,75 mmol/L (>11 mg/dL) II. Renal insufficiency: serum creatinine > 177 μmol/l (>2 mg/dl) III. Anemia: hemoglobin value of >20 g/l below the lower limit of normal or a hemoglobin value lower than 10g/dl.

   IV. Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET- CT (positron emission tomography) V. Clonal BM plasma cell percentage ≥60% VI. Involved: uninvolved serum free light chain ratio ≥100 VII. >1 focal lesion on MRI examination
2. Presence of measurable disease:

   I. Serum M-protein ≥ 0.5 g/dL or urine M-protein ≥ 200 mg/24 hours. II. Involved FLC (free light chain) level ≥ 10 mg/dl, provided sFLC (free light chain) ratio is abnormal.
3. R-ISS stage I33 (see appendix 2)
4. Standard gene expression pattern of isolated plasma cell based on SKY92 GEP assay
5. Must be ≥ 18 and ≤70 years at the time of signing the informed consent form.
6. Must be able to adhere to the study visit schedule and other protocol requirements in the investigator's opinion.
7. WHO (see Appendix 3) performance status 0-2 (WHO=2 is allowed only if caused by MM and not by co-morbid conditions).
8. Ability to understand and willingness to sign written informed consent. Signed informed consent must be obtained before any study specific procedure.
9. Suitable for high-dose melphalan and stem cell retransfusion.
10. Subjects must have adequate vascular access for leukapheresis

    .
11. Male or Female

Male participants:

A male participant must agree to use contraception during the intervention period and for at least 5 months after the last dose of isatuximab treatment and refrain from donating sperm during this period.

Female participants:

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

i) Not a Female of childbearing potential (FCBP), OR ii) A FCBP who must have a negative serum or urine pregnancy test with a sensitivity of at least 25 milliliter units (mIU)/mL within 28 days prior to and again within 24 hours prior to starting study medication and before each cycle of study treatment as well as day 21 of induction and experimental arm consolidation as well as every 28 days during all other cycles. If heavy menstruation appears or a menstruation is delayed, additional tests have to be performed. Participants must either commit to continue abstinence from heterosexual intercourse or apply a highly effective method of birth control during the intervention period and for at least 5 months after the last dose of isatuximab treatment Of note: contraception duration should take also into consideration any backbone therapy

All females:

Must understand the damages and hazards lenalidomide can cause to an unborn fetus and the necessary precautions associated with the use of lenalidomide.

Females of childbearing potential (FCBPs) must understand the need for effective contraception, without interruption. This should be 28 days before starting lenalidomide, isatuximab, throughout the entire duration of study and at least 5 months after the last dose of lenalidomide or isatuximab.

All female and male patients with fertile partners must adhere to the following recommendations:

I. If the female patients are permanently sterile or post-menopausal, they are considered to have no childbearing potential. Permanent sterilization methods include hysterectomy, bilateral salpingectomy. The postmenopausal state is defined as the absence of menstruation within 12 months without alternative medical reasons.

II. Female patients with fertility (and male patients with fertile partners) must agree to use an effective method of contraception (pearl index <1) throughout the study period and for 12 months thereafter.

III. According to the "Recommendations Related to Contraception and Pregnancy Tests in Clinical Trials" (Clinical Trial Facilitation Group, 2014-09-15), birth control methods considered to be very effective include:

* Combined (including estrogen and progesterone) hormonal contraception related to ovulation suppression*:

  * oral
  * In the vagina
  * Transdermal *Due to the increased risk of venous thromboembolism in subjects with multiple myeloma taking lenalidomide and dexamethasone, the use of combined oral contraceptive pills are not recommended and the method should be changed
* Progesterone-only hormone contraception associated with inhibition of ovulation*:

  * oral
  * Injectable
  * Implantable
* Intrauterine device (IUD)
* Intrauterine Hormone-releasing System (IUS)
* Vasectomized partner (with confirmed surgical success)
* Sexual abstinence (when consistent with the subject's usual lifestyle) IV. Investigational medicial product (IMP) may interact with hormonal contraceptives and may reduce the effectiveness of contraceptive methods V. Women using hormonal contraceptives should add a barrier method as a second form of contraception, because it is currently unknown whether lenalidomide, isatuximab, bortezomib or dexamethasone may reduce the effectiveness of hormonal contraceptives.

VI. Breast-feeding lenalidomide and its metabolites are excreted in human milk. It is unknown whether isatuximab is secreted in milk. A risk to the newborns/infants cannot be excluded. Breast-feeding should be discontinued during treatment with lenalidomide and isatuximab VII. Must adhere to regular pregnancy tests (at least every 21 days during induction and consolidation (experimental arm) and 28 days during maintenance and other therapy cycles, in case of irregular menstruation at least every two weeks, if heavy menstruation appears or menstruation is delayed, additional tests have to be performed).

VIII. Notify investigator if method of contraception is changed. IX. Notify investigator immediately in case of pregnancy

Male subjects must agree:

I. to use a condom during sexual contact with a pregnant female or a FCBP while taking lenalidomide or isatuximab, during any dose interruptions and for 5 months after the last dose of lenalidomide or isatuximab, II. Not donate semen or sperm while receiving lenalidomide, during dose interruptions and for at least 5 months after the last dose of lenalidomide and/or isatuximab.

III. Receive counseling about pregnancy precautions and the potential risks of fetal exposure to lenalidomide at a minimum of every 28 days l) All subjects must: I. Agree to abstain from donating blood while taking lenalidomide, during dose interruptions and for at least 5 months after the last dose of lenalidomide and/or Isatuximab.

II. Agree never to give lenalidomide to another person. III. Agree to return all unused lenalidomide capsules to the investigator (with exception of prescribed lenalidomide capsules) IV. Be aware that no more than a 28-day lenalidomide supply may be dispensed with each cycle of lenalidomide during induction and consolidation therapy and be prescribed during maintenance therapy.

Exclusion Criteria:

1. Direct Coombs test positive hemolytic anemia.
2. Involvement of the central nervous system (CNS).
3. History or presence of clinically relevant CNS pathology such as clinically relevant epilepsy, seizure, paresis, aphasia, stroke, subarachnoid hemorrhage or other CNS bleed, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
4. Subject with active or history of plasma cell leukemia, Waldenström's macroglobulinemia, POEMS syndrome or clinically significant amyloidosis.
5. Patients having nonsecretory MM.
6. Systemic AL amyloidosis (with exception of AL amyloidosis of BM).
7. Previous chemotherapy or radiotherapy during the past 5 years except local radiotherapy in case of local myeloma progression or benign diseases, such as nonmalignant thyroid diseases. (Note: patients may have received a cumulative dose of up to 320 mg of dexamethasone or equivalent as emergency therapy.) Previous therapy due to smouldering myeloma or a single dose of bortezomib may be acceptable. In this case the coordinating investigator or his deputy has to be consulted prior to inclusion.
8. Patients with any of the following laboratory abnormalities:

   I. Absolute neutrophil count (ANC) < 1,000/μL. II. Platelet count < 50,000/µL (Platelet transfusions are not permitted to improve platelet count one week prior to study inclusion.) III. Serum Creatinine Clearance (CrCl) < 30 mL/min/1,73m2. IV. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × upper limit of normal (ULN) (unless due to liver infiltration by myeloma cells), serum total bilirubin > 1.5 × ULN or > 3.0 mg/dL for subjects with documented Gilbert's syndrome.

   V. International ratio (INR) or partial thromboplastin time (PTT) > 1.5 × ULN, or history of Grade ≥ 2 hemorrhage within 30 days, or subject requires ongoing treatment with chronic, therapeutic dosing of anticoagulants (e.g. warfarin, low molecular weight heparin, or Factor Xa inhibitors).
9. Echocardiogram (ECHO) with left ventricular ejection fraction < 45%.
10. An inadequate pulmonary function defined as oxygen saturation (Sa02) < 92 % on room air
11. Known to be HIV+ or to have hepatitis A, B, or C active infection.

    Uncontrolled or active hepatitis B virus (HBV) infection: Patients with positive HBsAg and/or HBV DNA

    Of note:

    Patient can be eligible if anti-HBc immunoglobulin G (IgG) positive (with or without positive anti-HBs) but HBsAg and HBV DNA are negative.

    If anti-HBV therapy in relation with prior infection was started before initiation of IMP, the anti-HBV therapy and monitoring should continue throughout the study treatment period.

    Patients with negative HBsAg and positive HBV DNA observed during screening period will be evaluated by a specialist for start of anti-viral treatment: study treatment could be proposed if HBV DNA becomes negative and all the other study criteria are still met.

    Active HCV infection: positive HCV RNA and negative anti-HCV

    Of note:

    Patients with antiviral therapy for HCV started before initiation of IMP and positive HCV antibodies are eligible. The antiviral therapy for HCV should continue throughout the treatment period until seroconversion.

    Patients with positive anti-HCV and undetectable HCV RNA without antiviral therapy for HCV are eligible.
12. Subjects with prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years.
13. Subjects with severe polyneuropathy with accompanying pain
14. Hypersensitivity or allergy against any of the study drugs.
15. Contraindications against any of the study drugs as outlined in the Investigator brochure or equivalent.
16. Prisoners or subjects who are legally institutionalized, or those unwilling or unable to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
17. Participation in another interventional clinical trial during this trial or within 4 weeks before entry into this trial. There may be exceptions at the discretion of the (coordinating) investigator.
18. Active systemic infection and severe infections requiring treatment with a parenteral administration of antibiotics.
19. Any clinically significant, uncontrolled medical conditions that, in the Investigator's opinion, would expose the patient to excessive risk or may interfere with compliance or interpretation of the study results.
20. Hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Rate of minimal residual negativity combined with complete remission rate according to IMWG and EuroFlow criteria | Week 40 after start of induction therapy (18 weeks after randomization).
  Minimal Residual Disease (MRD) (less than 1 malignant plasma cell per 1 Mio bone marrow cells based on EuroFLow criteria) and complete remission rate (no paraprotein detectable, Immunfixation negative urine and serum) according to international myeloma working group (IMWG) criteria after high dose chemotherapy or 6 courses of IVRD (Isatuximab, Bortezomib, lenalidomide, Dexamethasone) (week 40)

SECONDARY OUTCOMES:
PFS | from inclusion till end of overall study
  to compare the two arms regarding Progression free survival (PFS) [ Time Frame: time from study inclusion to progression or death whichever comes first] from start of therapy till maximum of 5 years after start of trial
OS | From start to end of overall study
  to compare the two arms regarding Overall survival [ Time Frame: time from study inclusion) to death up to a maximum of 5 years
Toxicity | From start to end of overall study
  Number of adverse events in both arms, Toxicity during induction and maintenance with respect to adverse events of National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) grade >3 up to 5 years after start of treament
Response criteria | week 20, week 40, year 1, year 2
  Response according to IMWG criteria at week 20, 40, 1 year and 2 years after start of trial
Response criteria MRD | week 20, week 40, year 1, year 2
  Rate of MRD negativity (less than 10-5) at week 20, 40, 1 year and 2 years after start of trial
Quality of life (EORTC-5 questionnaire) | week 20, 40, year 1, year 2
  Quality of Life Assessment [based on EORTC-5 questionnaire) Time Frame: assessed at baseline, at week 20, 40, 1 year ) and 2 years after start of trial

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus Khandanpour, Prof. Dr., Principal Investigator — University Hospital Schleswig-Holstein, Campus Lübeck
Locations (6):
- Germany (6):
  - Heloisklinikum Berlin Buch GmbH, Berlin
  - Klinikum Bielefeld - Onkologie, Hämatologie, Paliativmedizin, Bielefeld
  - Universitätsklinikum Hamburg Eppendorf (UKE), Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Würzburg, Würzburg